CLINICAL TRIAL: NCT06022159
Title: Phase II Study Evaluating Pre-operative HYPOfractionated Radiation Therapy in Aged (≥ 70 Years) or "Fragile" (≥ 65 Years) Patients With Limb or Trunk Soft Tissue SARComa.
Brief Title: A Study to Evaluate Pre-operative HYPOfractionated Radiation Therapy in Aged (≥ 70 Years Old) or "Fragile" (≥ 65 Years) Patients With Limb or Trunk Soft Tissue SARComa.
Acronym: HYPOSARC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23 SARC 01
Record Dates: First submitted 2023-08-16; First posted 2023-09-01 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Soft Tissue Sarcoma
Keywords: Soft Tissue Sarcoma; Limb soft tissue SARComa; Trunk soft tissue SARComa; Aged population; "Fragile" population; hypofractionated radiation therapy
MeSH Terms: conditions — Sarcoma | interventions — Radiotherapy, Intensity-Modulated; Conservative Treatment

STUDY DESIGN:
Intervention Model Description: Radiation therapy followed by surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiation therapy followed by surgery (Experimental)
  Interventions: Radiation: Hypofractionated Radiation Therapy; Procedure: Conservative treatment

INTERVENTIONS:
Radiation: Hypofractionated Radiation Therapy — The Hypofractionated Intensity-Modulated Radiation Therapy will be delivered in 5 fractions of 6 Gy each on the Planning Target Volume (PTV). The total dose of 30 Gy will be administered in approximately 1 week.
  Other Names: Intensity-modulated radiation therapy (IMRT)
Procedure: Conservative treatment — A wide en bloc resection is required (amputation is excluded) while ensuring the best functional preservation. The surgical procedure will take place about 1,5 to 2 months after the end of the radiation therapy.

SUMMARY:
This is a phase II, multicenter, non-randomized study.

The main objective is to evaluate the treatment with hypofractionated radiation therapy in neo-adjuvant situations on wound healing in a population of aged patients (≥ 70 years old) or ≥ 65 years of age defined as "fragile" and treated for soft tissue sarcoma.

A maximum of 48 evaluable patients will be included in this study. The patients will receive an hypofractionated radiation therapy prior to conservative surgery.

Each patient will be followed for up to 3 years after the end of complete treatment (radiotherapy + surgery).

ELIGIBILITY:
Inclusion Criteria:

1. Patient with histologically confirmed soft tissue sarcoma of the limbs or trunk.
2. Indication for neo-adjuvant or adjuvant radiotherapy.
3. Patient aged ≥ 70 years with a performance status ECOG ≤ 2 and/or aged 65 to 70 years with an ECOG of 2 and identified by the investigator as "fragile".
4. Patient affiliated to a Social Health Insurance in France.
5. Patient able to participate and willing to give informed consent prior performance of any study-related procedures.

Exclusion Criteria:

1. Retroperitoneal, ORL and visceral sarcomas.
2. Previous radiotherapy in the area.
3. Metastatic disease.
4. Concomitant or sequential chemotherapy.
5. Patient requiring total surgery (amputation).
6. Other cancer under treatment.
7. Any condition or pathology contraindicating MRI.
8. Any psychological, familial, geographic or social situation, potentially preventing the provision of informed consent or compliance to study procedure.
9. Patients included in another therapeutic interventional trial.
10. Patient who has forfeited his/her freedom by administrative or legal award or who is under legal protection (curatorship and guardianship, protection of justice).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
The rate of patients free of major surgical complications as defined by O'Sullivan within 6 months of surgery. | 6 month for each patient

SECONDARY OUTCOMES:
Patients' disease-free survival defined as the time between the inclusion date and the occurrence of a carcinological event (local recurrence, distant metastasis) or death from any cause. | 3 years for each patient
Surgical complications evaluated according to NCI CTC AE V5 criteria. | 3 years for each patient
Wound disorders, such as partial necrosis and scar disunion, classified into four categories: severe, moderate, minor, absent. | 3 years for each patient
Healing time defined as the time between the date of surgery and the date of complete healing. | 3 years for each patient
Patients' quality of life evaluated using the EORTC questionnaire (QLQ-C30). | 3 years for each patient
Patients' quality of life evaluated using the EORTC questionnaire (QLQ-ELD14). | 3 years for each patient
Patient autonomy evaluated using the IADL (Instrumental Activities of Daily Living) questionnaire. | 3 years for each patient
Geriatric parameters evaluated using the G8 (Geriatric 8) questionnaire. | 3 years for each patient
Geriatric parameters evaluated using the G-CODE questionnaire. | 3 years for each patient
Toxicities of the radiation therapy evaluated according to NCI CTC AE V5 criteria and Radiation Therapy Oncology Group (RTOG) classification. | 3 years for each patient

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - Institut Bergonie, Bordeaux
  - Centre Oscar Lambret, Lille
  - Chu de Limoges, Limoges
  - Centre Leon Berard, Lyon
  - Institut Regional Du Cancer de Montpellier, Montpellier
  - Institut Curie, Paris
  - Chu de Poitiers, Poitiers
  - Institut de Cancerologie de L'Ouest, Saint-Herblain
  - Chu de Toulouse, Toulouse
  - IUCT-O, Toulouse
  - Institut Gustave Roussy, Villejuif